CLINICAL TRIAL: NCT05830253
Title: Free-living Monitoring of Parkinson's Disease Using Smart Objects: Towards Digital Medicine
Brief Title: Free-living Monitoring of Parkinson's Disease Using Smart Objects
Acronym: FREEDOM
Status: Completed | Type: Observational
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Dept. of Electronics, Informatics, Bioengineering, Politecnico di Milano, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 2574CE
Record Dates: First submitted 2023-03-08; First posted 2023-04-26 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Parkinson's disease, one of the most common neurodegenerative diseases of the central nervous system, presents motor symptoms, including tremor, rigidity, bradykinesia, and postural instability. Assessments of patients with Parkinson's disease are typically performed using clinical scales, compiled by the healthcare staff or by the patient. Although commonly used in clinical practice, they have some limitations, including the low temporal resolution of the scales, the low granularity of the scores and the possible low inter- and intra-operator reliability. The recent development of digital technologies has led to the creation of IoT (Internet of Things) devices capable of providing quantitative indicators, potentially useful for an accurate differential diagnosis, as well as for monitoring the effects of therapeutic interventions. The peculiarity of these systems is the ability to provide indicators not only during periodic visits to the clinic, but also the ability to remotely monitor the patient's daily life activities. In this scenario, this study wants to test the hypothesis that the IoT devices like smart-ink pens and insoles are usable options for monitoring patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuls
* Cognitive impairments
* Ability to independently sign the written informed consent

Exclusion Criteria:

* Unstable pharmacological treatment for Parkinson's Disease during the study
* Previous history of major neurological, vascular, musculoskeletal disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
System Usability Scale | 1-2 weeks
  Score ranges from 0 (no usability) to 100 (excellent usability)

SECONDARY OUTCOMES:
Movement Disordered Society - Unified Parkinson's Disease Rating Scale | Baseline
  Parkinson's Disease prognosis information. Score ranges from 0 (normal) to 199 (severe impairment).
Execution handwriting time | Baseline
  Time required to complete the handwriting task measured by the smart ink pen, in seconds
Execution handwriting time | 1-2 weeks
  Time required to complete the handwriting task measured by the smart ink pen, in seconds
Average handwriting force | Baseline
  The average exerted force during handwriting task measured by the smart ink pen, in arbitrary units
Average handwriting force | 1-2 weeks
  The average exerted force during handwriting task measured by the smart ink pen, in arbitrary units
Gait speed | Baseline
  Gait speed [cm/s] measured by sensorized insoles
Gait speed | 1-2 weeks
  Gait speed [cm/s] measured by sensorized insoles

CONTACTS AND LOCATIONS:
Locations (1):
- Istituti Clinici Scientifici Maugeri, Milan, Italy

IPD SHARING:
Plan to Share IPD: No